CLINICAL TRIAL: NCT03504163
Title: Phase II Study of Pembrolizumab (MK-3475) and Bacillus Calmette-Guérin (BCG) as First-Line Treatment for High-Risk T1 Non-Muscle- Invasive Bladder Cancer (NMIBC) and High- Grade Non-Muscle- Invasive Upper Tract Urothelial Cell Carcinoma (NMI-UTUCC)
Brief Title: Pembrolizumab (MK-3475) and Bacillus Calmette-Guérin (BCG) as First-Line Treatment for High-Risk T1 Non-Muscle-Invasive Bladder Cancer (NMIBC) and High-Grade Non-Muscle-Invasive Upper Tract Urothelial Carcinoma (NMI-UTUC)]
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-602
Record Dates: First submitted 2018-04-11; First posted 2018-04-20 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Bladder Cancer
Keywords: Pembrolizumab (MK-3475); Bacillus Calmette-Guérin (BCG); 17-602
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is a phase II trial of Pembrolizumab (MK-3475) in combination with Bacillus Calmette-Guérin (BCG) as first-line therapy in patients with high-risk T1 bladder cancer and also in an exploratory cohort of patients with high-grade NMI-UTUC.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Risk T1 Bladder Cancer Cohort (Experimental): Pts will receive pembrolizumab/MK-3475 after transurethral resection of bladder tumor/TURBT in comb w/BCG as initial therapy. Pembrolizumab (MK-3475) will be administered as a 400 mg IV infusion at 6-wk intervals for 9 doses over a 48-wk period, unless there is unacceptable toxicity or other reasons to discontinue treatment occur. Intravesical BCG therapy (TICE strain, 50 mg) will be given 1x-weekly for 6 consecutive wks as a standard induction course, followed by maintenance BCG consistent w/standard clinical practice. BCG will start on wk 3 after the first infusion of pembrolizumab (400 mg) to allow for initial priming of T cells to further enhance the effects of BCG treatment.
  Interventions: Drug: Pembrolizumab (MK-3475); Drug: Bacillus Calmette-Guérin (BCG)
- Exploratory cohort for high-grade non-muscle-invasive upper tract urothelial carcinoma (Experimental): Pts will receive pembrolizumab (MK-3475) administered after ureteroscopy/laser ablation in comb w/BCG as initial therapy. Pembrolizumab (MK-3475) will be administered as 400 mg IV infusion at 6-week intervals for 9 doses over a 48-week period, unless there is unacceptable toxicity or other reasons that would warrant the discontinuation of treatment. Pts will receive once-weekly BCG therapy (TICE strain, 50 mg) for 6 consecutive wks as a standard induction course administered through a percutaneous nephrostomy tube in antegrade fashion for patients with high-grade NMI-UTUC, consistent with standard clinical practice. BCG will start on wk 3 after the first infusion of pembrolizumab (400 mg) to allow for initial priming of T cells to further enhance the effects of BCG treatment.
  Interventions: Drug: Pembrolizumab (MK-3475); Drug: Bacillus Calmette-Guérin (BCG)

INTERVENTIONS:
Drug: Pembrolizumab (MK-3475) — Pembrolizumab (MK-3475) will be administered as a 400 mg intravenous (IV) infusion at 6- week intervals for 9 doses over a 48-week.
Drug: Bacillus Calmette-Guérin (BCG) — Intravesical BCG will be administrated once per week over a 6-week period as induction therapy, followed by maintenance BCG consistent with standard clinical practice

SUMMARY:
The purpose of this study is to find out the effectiveness of pembrolizumab in combination with BCG as a first line therapy for participants with high grade T1 bladder cancer who are at "high risk" for BCG alone to be ineffective and are seeking an alternative treatment option to radical cystectomy. There is biologic rationale for combining pembrolizumab and BCG as two distinct immunotherapies with possible additive or synergistic activity in urothelial cancer. The combination of pembrolizumab with BCG will also be evaluated in an exploratory cohort of patients with upper tract urothelial cancer.

DETAILED DESCRIPTION:
Patients will receive pembrolizumab (MK-3475) administered after TUR in combination with BCG as initial therapy. Pembrolizumab (MK-3475) will be administered as a 400 mg IV infusion at 6-week intervals (Q6W) for 9 doses over a 48 week period, unless there is unacceptable toxicity or other reasons that would warrant the discontinuation of treatment. Patients will receive once-weekly BCG therapy (TICE strain, 50 mg) for 6 consecutive weeks as a standard induction course, given as intravesical BCG for patients with T1 bladder cancer, and administered through a percutaneous nephrostomy tube in antegrade fashion for patients with high-grade NMI-UTUC, consistent with standard clinical practice. BCG will start on week 3 after the first infusion of pembrolizumab (400 mg) to allow for initial priming of T cells to further enhance the effects of BCG treatment. Initiation of induction BCG may be delayed (up to 14 days) if deemed clinically indicated by the treating physician due to side effects from TURBT or ureteroscopy and with permission from the Principal Investigator (PI).

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Histologically confirmed urothelial cancer by TURBT performed at MSK for patients in the T1 bladder cancer cohort or by high-grade cytology/biopsy by ureteroscopy performed at MSK for patients in the NMI-UTUC cohort.
* TURBT within 8 weeks of protocol entry with complete resection of all papillary lesions for patients in the T1 bladder cancer cohort and ureteroscopy within 8 weeks of protocol entry with complete ablation of all papillary lesions with ureteroscopy or through antegrade percutaneous access for patients in the NMI-UTUC cohort..
* Patients in the T1 bladder cancer cohort must have high risk, BCG-naïve non-muscle-invasive urothelial cancer defined as having one of the following disease states:

  * T1 on restaging biopsy, plus CIS
  * Multiple (≥ 1) T1 recurrences, plus CIS
  * Multifocal T1 plus CIS
  * T1b (extensive/deep invasion into lamina propria) plus CIS
  * Lymphovascular invasion plus CIS
  * T1 with variant histology: including micropapillary, nested variant, poorly differentiated, squamous, and glandular differentiation (the presence of variant histology will be based on MSKCC review), plus CIS.
  * T1 with urothelial carcinoma of prostatic urethra (Ta, Tis, or T1 within prostatic urethra), plus CIS
  * Large (≥3 cm) T1 tumor, plus CIS
* Patients in the NMI-UTUC cohort must have high risk, BCG naïve NMI-UTUC, defined by having one of the following disease states:

  * Histologic confirmed ureteroscopic biopsy with clinical stage Tis (also known as CIS), Ta, or T1 disease in the renal pelvis. Concomitant ureteral disease will be allowed if completely treated endoscopically.
  * Clinical stage Tis confirmed by a positive high-grade selective cytology, coupled with ureteroscopic evaluation, confirming only flat eryethematous lesions and the absence of papillary tumors.
  * Must not have received prior treatment with percutaneous BCG to the involved renal unit, but prior intravesical BCG for bladder cancer is acceptable.
* Patients must have cross sectional imaging (CT or MRI urogram) within 3 months of protocol entry demonstrating no evidence of metastasis or radiographic evidence of muscle invasive disease.
* Patient refusal of cystectomy and bilateral pelvic lymphadenectomy for the T1 bladder cancer cohort, or refusal of radical nephroureterectomy for NMI-UTUC cohort.
* No prior intravesical BCG therapy for patients in the T1 bladder cancer cohort.
* No prior radiation therapy for bladder cancer for patients in the T1 bladder cancer cohort. Prior radiation therapy for prostate cancer is allowed.
* ECOG performance status of 0 or 1.
* Age ≥ 18 years.
* Female subjects of childbearing potential must be willing to use 2 methods of birth control, be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of the study medication (reference section 9.5.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for >1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Patients must not have other invasive malignancies within the past 5 years (with the exception of non-melanoma skin cancers, localized prostate cancer, and CIS of the cervix).
* Required initial laboratory values:

  * Absolute neutrophil count ≥ 1.5 x 10^9/L
  * Platelets ≥ 100 x 10^9/L
  * Hemoglobin ≥ 9 g/dL
  * Bilirubin ≤ 1.5 times the upper limit of normal (x ULN)
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 x ULN
  * Calculated creatinine clearance ≥ 30 using the CKD-Epi formula

Exclusion Criteria:

* Current or History of muscle invasive bladder cancer or prostatic stromal invasion.
* Unstable angina
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction within 6 months
* History of stroke within 6 months
* Evidence of bleeding diathesis or coagulopathy
* Presence of any systemic metastases (i.e, nodal, visceral, or central nervous system)
* Major surgical procedure (other than TURBT or ureteroscopy) within 28 days prior to the study
* Pregnant (positive pregnancy test) or lactating
* Serious, non-healing wound, ulcer, or bone fracture
* Inability to comply with study and/or follow-up procedures
* Prior therapy with an anti-PD-1 agent, anti-PD-L1 agent, or other inhibitory or stimulatory agent oriented towards a T-cell receptor
* Active infection requiring systemic therapy
* Known history of human immunodeficiency virus (HIV)
* Known active Hepatitis B or Hepatitis C
* Received live attenuated vaccines within 30 days prior to start of study treatment. Patients must also agree to avoid live attenuated vaccines during study treatment.
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic or immunosuppressive agents. Subjects with vitiligo, diabetes Type I, or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators, inhaled steroids, or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjøgren's syndrome will not be excluded from the study.
* Known contraindications to BCG, defined as one of the following:

  * History of systemic hypersensitivity reaction or history of febrile systemic BCG reaction
  * Febrile illness or persistent gross hematuria
  * Active tuberculosis
  * Immunosuppression due to congenital or acquired immune deficiency, concurrent immune suppressive disease, systemic cancer therapy, or chronic immunosuppressive therapy other than topical or inhaled corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who are disease-free | 6 months
  The primary objective for the high-risk T1 bladder cohort is to estimate the proportion of patients who remain free from high-grade recurrence (by urine cytology, cystoscopy ± biopsy) at 6 months from the start of treatment with pembrolizumab (MK-3475) and BCG

SECONDARY OUTCOMES:
The proportion of patients who remain free from high-grade recurrence | 6 months
  Determine the proportion of patients who remain free from high-grade recurrence (by urine cytology, cystoscopy ± biopsy) at 12 months from the start of treatment with pembrolizumab (MK-3475) and BCG

CONTACTS AND LOCATIONS:
Overall Officials: Gopakumar Iyer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All protocol activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (All protocol activities), Commack, New York
  - Memorial Sloan Kettering West Harrison (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm